CLINICAL TRIAL: NCT01362829
Title: Outcome Predictors in Patients With Severe Sepsis and Optimized Central Venous Oxygen Saturation
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Yu, Chong-Jen/MD, PhD, National Taiwan University Hospital
Other Study IDs: 200907064R; 098014-3 (Other: Far Eastern Memorial Hospital)
Record Dates: First submitted 2011-05-24; First posted 2011-05-30 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-05

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For each patient enrolled, 10mL blood is collected in EDTA-coated tube, which will be used for plasma separation and for peripheral blood mononuclear cell collection.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with severe sepsis: Patients who are admitted to medical ICU with severe sepsis
  Interventions: Other: Determined by intended physician

INTERVENTIONS:
Other: Determined by intended physician — We perform a prospective observational study. All the treatment for the patients are determined by intended physicians.

SUMMARY:
The investigators perform a prospective observation study to search for the outcome predictors (ScvO2 and lactate) in patients with severe sepsis after admission to ICU.

DETAILED DESCRIPTION:
Early goal-directed therapy in patients with severe sepsis or septic shock was found to provide survival benefit.It was thought that early optimization of ScvO2 within 6 hours in emergency department brought survival benefit to patients of septic shock or severe sepsis.On the other hand, early lactate clearance is associated with improved outcome in patients with severe sepsis or septic shock. In patients with severe sepsis and septic shock, those with low lactate clearance had poor prognosis, despite optimization of ScvO2. It is unknown if ScvO2 could still guide hemodynamic resuscitation after admission into ICU. The investigators perform a prospective observation study to see the correlation between ScvO2 and clinical outcome (including organ failure, disease severity, and survival) and the correlation between lactate and clinical outcome. Furthermore, if ScvO2 >= 70% is still of prognostic significance in ICU, we will investigate the outcome in patients with high ScvO2 and high serum lactate levels, and to evaluate the clinical features of this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are admitted to medical intensive care units with severe sepsis or septic shock

Exclusion Criteria:

* Patients would be excluded if they have any one of the exclusion criteria, *including pregnancy

  * presence of acute cerebral vascular attack
  * acute cardiogenic lung edema
  * status asthmatics
  * cardiac dysrhythmia as the primary diagnosis
  * massive gastrointestinal bleeding
  * epileptics
  * drug overdose
  * requirement of immediate surgery
  * hematologic malignancies
  * febrile neutropenia
  * treatment with immunosuppressive agents before admission
  * advanced malignancy and poor pre-admission performance status
  * with inevitable short-term mortality or morbidity
  * HIV infection
  * refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are admitted to medical intensive care units due to severe sepsis or septic shock
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
28-day Mortality | 28 days
  Record 28-day all-cause mortality in each population (low ScvO2, high ScvO2 and low serum lactate, high ScvO2 and high serum lactate)

SECONDARY OUTCOMES:
In-Hospital Mortality | 2 months
  Participants will be followed for the duration of hospital stay, an expected average of 2 months
Severity of organ failure | 1 week
  To evaluate the development of ARDS/ALI, AKI, and the record the SOFA score

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Jen Yu, MD, PhD, Principal Investigator — National Taiwan University Hospital; Hou-Tai Chang, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (2):
- Taiwan (2):
  - Far Eastern Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei